CLINICAL TRIAL: NCT02559830
Title: A Phase I/II Clinical Trial of Lentiviral Hematopoietic Stem Cell Gene Therapy for Treatment of Developed Metachromatic Leukodystrophy and Adrenoleukodystrophy
Brief Title: Autologous Hematopoietic Stem Cell Gene Therapy for Metachromatic Leukodystrophy and Adrenoleukodystrophy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Collaborators: Shenzhen University (Other); Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChiCTR-OPC-15005802
Record Dates: First submitted 2015-08-12; First posted 2015-09-24 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2016-09

CONDITIONS: Metachromatic Leukodystrophy; Adrenoleukodystrophy
MeSH Terms: conditions — Leukodystrophy, Metachromatic; Adrenoleukodystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- transduced CD34+ hematopoietic stem cell (Experimental): Transplantation of autologous CD34+ hematopoietic stem cells transduced with ARSA/ABCD1 encoding lentiviral vector. Dosage: 2x10^6/Kg （Minimum）to 20x10^6/Kg （Maximum） transduced CD34+ cells at bedside for infusion
  Interventions: Genetic: transduced CD34+ hematopoietic stem cell

INTERVENTIONS:
Genetic: transduced CD34+ hematopoietic stem cell — Autologous hematopoietic stem cells (HSCs) collected from the mobilized peripheral blood and transduced ex vivo with a Lentiviral vector encoding the human ARSA(for MLD)/ABCD1(for ALD) cDNA（complementary DNA）. Dose: ≥ 2x10^6 transduced CD34+ cells/Kg (maximum 20x10^6) at bedside for infusion.

SUMMARY:
Evaluating the safety and efficacy of Lentiviral Hematopoietic Stem Cell Gene Therapy for advanced stage of Metachromatic Leukodystrophy and adrenoleukodystrophy.

DETAILED DESCRIPTION:
This is a phase I/II protocol aiming at the assessment of the safety and efficacy of arylsulfatase A（ARSA) / adenosine-triphosphate-binding cassette, sub-family D (ABCD1) gene transfer into hematopoietic stem/progenitor cells for the treatment of metachromatic leukodystrophy/adrenoleukodystrophy.

Metachromatic Leukodystrophy (MLD) is an autosomal recessive Lysosomal Storage Disorder (LSD) characterized by severe and progressive dysmyelination affecting the central and peripheral nervous system. Adrenoleukodystrophy (also known as X-linked adrenoleukodystrophy, ALD, X-ALD), a disorder of peroxisomal fatty acid beta oxidation which results in the accumulation of very-long chain fatty acids (VLCFA) in tissues throughout the body, is caused by mutations in ABCD1.Both diseases are characterized by progressive neurodegenerative decline, leading to a devastating state without treatment.

Hematopoietic cell transplantation (HCT) is ineffective in ameliorating patients' phenotype or delaying disease evolution in many patients. No evidences of efficacy of enzyme replacement strategies are available at the moment. Transplantation of genetically corrected autologous hematopoietic stem cells (HSC) could represent a novel and potentially efficacious treatment for MLD/ALD patients.

Recently, an Italian group conducted a gene therapy clinical trial based on autologous HSC and advanced generation lentiviral vectors (LV) for patients affected by the most severe, early onset forms of the disease (ClinicalTrials.gov Identifier:

NCT01560182).The safety and efficacy of this gene therapy approach in MLD patients was evaluated.During 3 years of follow-up, they reported multilineage ARSA expression and ability to prevent and correct neurological disease manifestations.However, only pre-symptomatic late infantile/Pre- or early-symptomatic early juvenile patients were recruited into the trial. In most cases, MLD/ALD patients tend to be diagnosed at an advanced stage, missing the best timing of curable HSC intervention. In our study, we intend to recruit symptomatic patients for transduced cluster of differentiation 34 positive (CD34+) HSC treatment. In the treated patients, we will study the short-term and long-term safety of the administration of the autologous transduced HSC, their long-term engraftment, the expression of vector-derived ARSA/ABCD1, and the ability of the transduced cells to provide a clinical benefit to the patients. The treated patients will be followed for 3 years and thereafter monitored for the safety of gene therapy for additional 5 years. If successful, this study will provide key results on the safety and efficacy of gene therapy for MLD/ALD patients.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria For MLD:

1. Confirmed diagnosis as MLD by ARSA genetic diagnosis, MRI（Magnetic Resonance Imaging）and low ARSA A activity (below 20% of normal level);
2. The patient' symptoms and lesions have not been developed to the end stage of MLD.
3. age < 16.0 years at symptom onset

Inclusion Criteria For ALD:

1. Confirmed diagnosis as ALD by ABCD1 genetic diagnosis, abnormal MRI imaging, abnormal high level of very long chain fatty acid (VLCFA) and adrenocorticotropic hormone (ACTH);
2. The patient' symptoms and lesions have not been developed to the end stage of ALD.
3. age < 16.0 years at symptom onset

Exclusion Criteria:

Exclusion Criteria For MLD：

1. At a pre-symptomatic stage of of MLD;
2. ARSA activity >50% compared to healthy individuals;
3. End stage of MLD;
4. Other complications, ie. Cancer;
5. human immunodeficiency virus（HIV） RNA and/or hepatitis C virus RNA and/or hepatitis B virus DNA positive patients;
6. Patients who underwent allogenic hematopoietic stem cell transplantation with evidence of residual cells of donor origin.
7. Serious organ dysfunction;
8. were enrolled in other clinical trials in the 6 months prior to screening;
9. had any other concern that hampered the compliance or safety as judged by the investigator;
10. Adult

Exclusion Criteria For ALD:

1. No evidence of brain lesions;
2. Normal level of VLCFAs in blood;
3. End stage of ALD;
4. Other complications, ie. Cancer;
5. human immunodeficiency virus（HIV） RNA and/or hepatitis C virus RNA and/or hepatitis B virus DNA positive patients;
6. Patients who underwent allogenic hematopoietic stem cell transplantation with evidence of residual cells of donor origin.
7. Serious organ dysfunction;
8. were enrolled in other clinical trials in the 6 months prior to screening;
9. had any other concern that hampered the compliance or safety as judged by the investigator;
10. Adult

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
The short-term safety and tolerability after hematopoietic stem cell transplanation | 2 months
  The absence of engraftment failure or delayed hematopoietic reconstitution (prolonged aplasia), defined as Absolute Neutrophil Count (ANC)<500/μl with no evidence of Bone Marrow recovery, requiring cellular back-up administration.
Incidence of Treatment-Emergent Adverse Events(For MLD) | 72 hours
  It will be evaluated on the basis of adverse events reporting and monitoring of the systemic reactions to cell infusion (fever, tachycardia, nausea and vomiting, joint pain, skin rash).
Incidence of Treatment-Emergent Adverse Events(For ALD) | 72 hours
  It will be evaluated on the basis of adverse events reporting and monitoring of the systemic reactions to cell infusion (fever, tachycardia, nausea and vomiting, joint pain, skin rash).
The long-term safety safety after hematopoietic stem cell transplanation | up to 8 years
  The absence of adverse affects in the long-term follow-up of HSCGT-treated patients, like hematopoietic system disease.

SECONDARY OUTCOMES:
ARSA activity for MLD | up to 8 years
  Before and after transplantation 1/2 year, 1 year, 3 years, 5 years, and 8 years (all time points are between plus or minus 0.5 years), residual ARSA activity (nmol/mg Prot/hr) measured in peripheral blood mononuclear cell (PBMC) and/or bone marrow progenitors will be tested (For MLD).
VLCFA level for ALD | up to 8 years
  Before and after transplantation 1/2 year, 1 year, 3 years, 5 years, and 8 years (all time points are between plus or minus 0.5 years), very long chain fatty acid(VLCFA) level ( C22,C24,C26 ,nmol/ml; C24/C22; C26/C22) in plasma will be measured (For ALD).
Magnetic Resonance imaging (MRI) score | up to 8 years
  Before and after transplantation 1/2 year, 1 year, 3 years, 5 years, and 8 years (all time points are between plus or minus 0.5 years), a detailed demerit scoring (0-34 points) developed by Dr. Loes will be performed in determining the extent of myelin injury in brain (eg, very early stage = MRI score 1-3; early stage = MRI score 4-8; late stage = MRI score 9-13; very late stage = MRI score greater than 13).
Functional independence measure (FIM) score | up to 8 years
  Before and after transplantation 1/2 year, 1 year, 3 years, 5 years, and 8 years (all time points are between plus or minus 0.5 years), a detailed FIM scores will be performed in determining the affect that neurodegeneration impair patients' independence for self-care.
Vector copy number (VCN) | up to 8 years
  Before and after transplantation 1/2 year , 1 year, 3 years, 5 years, and 8 years (all time points are between plus or minus 0.5 years), PBMCs from periheral blood will be seperated and DNA will be extracted, the VCN per cells will be investigated according to previosu publications by Biffi et al (Science,2013) .
Genomic lentiviral integration sites (Optional) | up to 8 years
  Before and after transplantation 1/2 year , 1 year, 3 years, 5 years, and 8 years (all time points are between plus or minus 0.5 years), peripheral blood mononuclear cell (PBMCs) from periheral blood will be seperated and DNA will be extracted, genomic lentiviral integration sites will be investigated according to previosu publications by Biffi etal (Science,2013) .

CONTACTS AND LOCATIONS:
Overall Officials: Qizhou Lian, M.D.,Ph.D., Principal Investigator — The University of Hong Kong; Jiacai Zhuo, Principal Investigator — Shenzhen Second People's Hospital; Xin Du, M.D.,Ph.D., Principal Investigator — Shenzhen Second People's Hospital; Hua Jiang, M.D,Ph.D, Principal Investigator — Guangzhou Women and Children's Medical Center; GuangFu Chen, M.D.,Ph.D, Principal Investigator — Shenzhen Second People's Hospital
Locations (1):
- Shenzhen Second People's Hospital, The First Affiliated Hospital of Shenzhen University, Shenzhen, Guangdong, China

REFERENCES:
- [Result] Cartier N, Hacein-Bey-Abina S, Bartholomae CC, Veres G, Schmidt M, Kutschera I, Vidaud M, Abel U, Dal-Cortivo L, Caccavelli L, Mahlaoui N, Kiermer V, Mittelstaedt D, Bellesme C, Lahlou N, Lefrere F, Blanche S, Audit M, Payen E, Leboulch P, l'Homme B, Bougneres P, Von Kalle C, Fischer A, Cavazzana-Calvo M, Aubourg P. Hematopoietic stem cell gene therapy with a lentiviral vector in X-linked adrenoleukodystrophy. Science. 2009 Nov 6;326(5954):818-23. doi: 10.1126/science.1171242. PMID 19892975
- [Result] Biffi A, Montini E, Lorioli L, Cesani M, Fumagalli F, Plati T, Baldoli C, Martino S, Calabria A, Canale S, Benedicenti F, Vallanti G, Biasco L, Leo S, Kabbara N, Zanetti G, Rizzo WB, Mehta NA, Cicalese MP, Casiraghi M, Boelens JJ, Del Carro U, Dow DJ, Schmidt M, Assanelli A, Neduva V, Di Serio C, Stupka E, Gardner J, von Kalle C, Bordignon C, Ciceri F, Rovelli A, Roncarolo MG, Aiuti A, Sessa M, Naldini L. Lentiviral hematopoietic stem cell gene therapy benefits metachromatic leukodystrophy. Science. 2013 Aug 23;341(6148):1233158. doi: 10.1126/science.1233158. Epub 2013 Jul 11. PMID 23845948
- [Result] Consiglio A, Quattrini A, Martino S, Bensadoun JC, Dolcetta D, Trojani A, Benaglia G, Marchesini S, Cestari V, Oliverio A, Bordignon C, Naldini L. In vivo gene therapy of metachromatic leukodystrophy by lentiviral vectors: correction of neuropathology and protection against learning impairments in affected mice. Nat Med. 2001 Mar;7(3):310-6. doi: 10.1038/85454. PMID 11231629
- [Result] Matzner U, Schestag F, Hartmann D, Lullmann-Rauch R, D'Hooge R, De Deyn PP, Gieselmann V. Bone marrow stem cell gene therapy of arylsulfatase A-deficient mice, using an arylsulfatase A mutant that is hypersecreted from retrovirally transduced donor-type cells. Hum Gene Ther. 2001 Jun 10;12(9):1021-33. doi: 10.1089/104303401750214258. PMID 11399225
- [Result] Patil SA, Maegawa GH. Developing therapeutic approaches for metachromatic leukodystrophy. Drug Des Devel Ther. 2013 Aug 8;7:729-45. doi: 10.2147/DDDT.S15467. eCollection 2013. PMID 23966770